CLINICAL TRIAL: NCT00004498
Title: Phase I Study of Adenoviral Vector Mediated Gene Transfer for Ornithine Transcarbamylase in Adults With Partial Ornithine Transcarbamylase Deficiency
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/14290; UPSM-FDR001529
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2000-02

CONDITIONS: Ornithine Transcarbamylase Deficiency Disease
Keywords: genetic diseases and dysmorphic syndromes; inborn errors of metabolism; ornithine transcarbamylase deficiency; rare disease; urea cycle disorder
MeSH Terms: conditions — Ornithine Carbamoyltransferase Deficiency Disease; Genetic Diseases, Inborn; Metabolism, Inborn Errors; Rare Diseases; Urea Cycle Disorders, Inborn

INTERVENTIONS:
Genetic: Adenoviral Vector-Mediated Gene Transfer

SUMMARY:
OBJECTIVES:

I. Determine the safety, feasibility, and potential efficacy of intravascular adenoviral vector mediated gene transfer in the liver in adults with partial ornithine transcarbamylase deficiency.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a dose escalation study. Patients undergo a femoral arterial placement of a hepatic intraarterial catheter. Patients then receive adenoviral vector mediated gene transfer intravascularly over 30 minutes.

Cohorts of 3 patients each receive escalating doses of adenoviral vector until the maximum tolerated dose is determined.

Patients are followed at 3, 5, 7, 8, 15, and 29 days, at 2 months, and then every 3 months thereafter.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of partial ornithine transcarbamylase deficiency Female heterozygote with abnormal allopurinol challenge or underlying defect in either N15 urea or N15 glutamine OR Male with childhood/adulthood onset OR Family history of 2 affected children
* Stable for at least 1 month prior to study
* Plasma ammonium levels less than 50 micromoles

--Prior/Concurrent Therapy--

* Concurrent alternate pathway therapy to control hyperammonemia allowed

--Patient Characteristics--

* Hepatic: No history of liver disease
* Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No high level of neutralizing antibodies to the adenovirus

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 1998-07; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Steven E. Raper, Study Chair — University of Pennsylvania